CLINICAL TRIAL: NCT02401490
Title: Albumin Infusion Effects in Mortality in Patients With Cirrhosis and Hepatic Encephalopathy
Acronym: BETA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BETA; 2014-004809-33 (EudraCT Number)
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hepatic Encephalopathy; Cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Human albumin (Active Comparator): human albumin in the 24-48 hours after the hospitalization and at 48+/- 24 hours after the first dose.
  Interventions: Drug: Human albumin
- placebo (Placebo Comparator): saline serum 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Human albumin — 1.5gr/Kg/day at least in the 24-48 hours after the hospitalization and 1.0 gr/Kg/day at 72 hours after the first dose.
  Arms: Human albumin
Drug: Placebo
  Arms: placebo

SUMMARY:
To assess whether albumin administration after an episode of hepatic encephalopathy (≥ grade II) improves survival at 90 days (mortality endpoint treated as a composite endpoint death and/ or liver transplantation).

DETAILED DESCRIPTION:
To evaluate whether albumin administration after an episode of hepatic encephalopathy (≥ grade II) improves survival at 30, 90 and 180 days.

* to evaluate the effects of albumin on hepatic encephalopathy recurrence during the study period.
* To analyze whether albumin administration reduces hospitalization requirement.
* To study the effects of albumin on circulatory dysfunction index (mean arterial pressure, renal function, plasma vasopressor hormones).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years.
2. Liver cirrhosis defined by previous clinical data or liver biopsy.
3. Presence of an episode of acute hepatic encephalopathy of grade> 2.
4. Sign the informed consent

Exclusion Criteria:

1. Pregnant or breast-feeding.
2. Terminal illness.
3. Presence of Acute-on-chronic liver failure.
4. Needing for intensive support measures.
5. Active gastrointestinal bleeding.
6. neurological or psychiatric comorbidity that hinders the assessment of hepatic encephalopathy.
7. Clinical situations in which it is contraindicated to administer intravenous albumin.
8. MELD score less than 15 or greater than 25 at the time of inclusion
9. Any medical condition previous to patient inclusion in the study involving administration of albumin during a previous 7 day period.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Survival at 90 days. (The mortality endpoint is treated as a composite endpoint mortality and / or liver transplantation). | 90 days

SECONDARY OUTCOMES:
Survival at 180 days. | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: German Soriano, Principal Investigator — Hospital de la Santa creu i Sant Pau - Barcelona; Jordi Sanchez, Principal Investigator — Corporació Sanitària Parc Taulí, Sabadell; Helena Masnou, Principal Investigator — Hospital Universitari Germans Trias i Pujol, Badalona; Núria Cañete, Principal Investigator — Hospital del Mar; Marta Martín, Principal Investigator — Hospital de Sant Joan Despí Moisès Broggi, Sant Joan Despí; Elsa Solà, Principal Investigator — Hospital Clinic of Barcelona
Locations (7):
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan Despí, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona